CLINICAL TRIAL: NCT03703180
Title: Vision Assessment With the qCSF Method in Healthy Controls and MS: Investigating the Association Between Optical Coherence Tomography (OCT) and qCSF Dynamics Over Two Years and Set-up of a Representative Normative Data-set
Brief Title: Vision Assessment With the Quick Contrast Sensitivity Function (qCSF) Method in Healthy Controls and MS
Acronym: VICTOR2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: inims-victor2
Record Dates: First submitted 2018-10-04; First posted 2018-10-11 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MS: representative cohort of relapsing-remitting MS (n=50) and progressive MS patients (n=50) over the typical age range of 18-65. During two years of follow-up the integrity and function of the visual system will be observed annually with optical coherence tomography, high and low contrast visual acuity and a vision related quality of life questionnaire.
- Controls: Age and Gender matched healthy controls (n=100) will undergo the same assessments as the MS cohort to build up a representative normative dataset.

SUMMARY:
Victor2 is an observational cohort study over two years and is designed to investigate longitudinal changes of visual impairment in multiple sclerosis (MS). The investigators aim to recruit patients in the relapsing-remitting phase of the disease (n=50) as well as progressive MS patients (n=50). Both cohorts will be compared with age and gender matched healthy controls (HC). All participants undergo yearly clinical assessments including standard charts for visual acuity (Sloan, Snellen), a new computer adaptive test measuring the complete contrast sensitive function (CSF), optical coherence tomography and a vision related quality of life questionnaire (NEI-VFQ). The study aims to validate and extend previous finding from a cross-sectional study which found a better association between CSF and NEI-VFQ than for standard charts. Moreover, the study is designed to proof also a better association with anterior visual system integrity as assessed with OCT.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria relapsing-remitting MS

* Relapsing-remitting MS
* Expanded Disability Status Scale (EDSS) Score between 0 and 6.0
* No other major neurological or psychiatric disorder (such as major depression or schizophrenia)
* Age 18 - 65 years

Inclusion criteria progressiveMS

* Primary or Secondary-progressive MS according to the revised McDonald criteria
* Expanded Disability Status Scale (EDSS) Score between 3.0 and 6.0
* No relapse in the last 12 months
* No other major neurological or psychiatric disorder (such as major depression or schizophrenia)
* Age 18 - 65 years

Exclusion Criteria:

* Cataract and other major ophthalmological diseases (e.g. Uveitis, Glaucoma)
* Hyperopia > 5 dpt, Myopia > -7 dpt, Astigmatisms > 3 dpt
* Neuromyelitis optica spectrum diseases

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: representative longitudinal cohort including the complete spectrum of disease course
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-29 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between ganglion cell / inner plexiform layer (GCIPL) thickness loss and area under the log CSF curve change over two years | 2 years
  GCIPL thickness represents anterior visual system integrity on neuronal level and its change over two years will be correlated with the change of the CSF

SECONDARY OUTCOMES:
Correlation between retinal nerve fibre layer (RNFL) thickness loss and area under the log CSF curve change over two years | 2 years
  To correlate anterior visual system integrity with contrast vision assessed with the CSF
Longitudinal correlation between visual quality of life and contrast vision | 2 years
  To correlate Quality of life scores from the national eye institute visual functioning questionnaire questionnaire with contrast vision assessed with the CSF

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Patrick Stellmann, MD, Principal Investigator — Institute of Neuroimmunology and MS
Locations (1):
- Institute of Neuroimmunology and MS, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous data will be available after study completion.